CLINICAL TRIAL: NCT03095443
Title: Decreasing Delirium Through Music
Acronym: DDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Regenstrief Institute, Inc. (Other)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1608887741
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Delirium
Keywords: Delirium; Critical Illness; Music Therapy
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Music (Experimental): Receives personalized playlist twice a day.
  Interventions: Other: Music Therapy - Personalized Playlist
- Non Personalized Music (Active Comparator): Receives standardized low beats per minute playlist twice a day.
  Interventions: Other: Music Therapy - Standard Playlist
- Attention Control (Active Comparator): Receives audio-book twice a day.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Music Therapy - Personalized Playlist — Participant receives personalized playlist.
  Arms: Personalized Music
Other: Music Therapy - Standard Playlist — Participant receives a standard low beats per minute playlist.
  Arms: Non Personalized Music
Other: Attention Control — Participant receives an audio-book.
  Arms: Attention Control

SUMMARY:
DDM is a study designed to Test the efficacy of personalized music therapy in reducing delirium incidence and severity among patients admitted to the Intensive Care Unit.

DETAILED DESCRIPTION:
Over 1 million adults are admitted to the intensive care unit and placed on mechanical ventilation on an annual basis. Intravenous sedatives and analgesics are commonly administered to these patients to reduce pain and anxiety. While the recent reduction in benzodiazepine usage has helped reduced ICU-related acute brain dysfunction (delirium), up to 80% of ventilated patients still develop acute brain failure. This is characterized by disturbance of consciousness with reduced ability to focus, sustain or shift attention, occurring over a short period of time and fluctuating over the course of a day.

Acute brain dysfunction has both short-term and long-term health impacts. It is associated with increased hospital length of stay, increased in-hospital mortality and post-discharge mortality as well increased health-care costs. Patients who experience delirium are at greater risk for post-discharge institutionalization and newly acquired cognitive impairment similar to dementia.

Despite the prevalence and morbidity associated with delirium, there is a scarcity of effective pharmacological and non-pharmacological interventions to prevent and treat this condition. While music therapy has shown to reduce anxiety and stress in cancer and dementia patients, these studies were performed outside the intensive care unit. It is hypothesized that music lowers inflammatory mediators such as cytokines and cortisol. Delirium pathophysiology similar to anxiety has a strong inflammatory component with excess of pro-inflammatory cytokines such as interleukins 1, 6, and 8. Given the beneficial effects of music in reducing inflammatory mediators, it stands to reason that such intervention will have a beneficial impact on reducing delirium.

The investigators propose a randomized, three-group (personalized music intervention versus generic music intervention versus attention control) trial to test the feasibility and efficacy of music therapy in reducing delirium incidence, duration, and severity among critically ill patients in the ICU.

Our study focuses on the effect of music therapy on the incidence and severity of delirium in the intensive care unit at a large urban academic health center.

The investigators hypothesize that music therapy will lead to reduced levels of anxiety, delirium and need for sedating medications, leading to shorter hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* English speaking
* admitted to the intensive care unit (medical or surgical)
* receiving mechanical ventilation

Exclusion Criteria:

* history of dementia
* psychiatric illness which is not well controlled
* alcohol withdrawal symptoms/concern for withdrawal
* suspected or confirmed drug intoxication/overdose
* traumatic brain injury
* hearing or vision impairment including legal blindness
* aphasic stroke
* coma after cardiac arrest/hypothermia protocol
* pregnant or nursing
* prisoners
* patients enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | Date of study enrollment through discharge from ICU, or date of study enrollment up to 28 days
  the number of participants approached and their rates of consent
Intervention adherence | Date of study enrollment through discharge from ICU, or date of study enrollment up to 28 days
  number of listening sessions completed per patient
Participant retention | Date of study enrollment through discharge from ICU, or date of study enrollment up to 28 days
  Number of patients who complete the study.

SECONDARY OUTCOMES:
Estimate the potential effect size | Date of study enrollment through discharge from ICU, or date of study enrollment up to 28 days
  Patient-preferred music association with reducing delirium incidence as measured by CAM-ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan SH, Wang S, Harrawood A, Martinez S, Heiderscheit A, Chlan L, Perkins AJ, Tu W, Boustani M, Khan B. Decreasing Delirium through Music (DDM) in critically ill, mechanically ventilated patients in the intensive care unit: study protocol for a pilot randomized controlled trial. Trials. 2017 Nov 29;18(1):574. doi: 10.1186/s13063-017-2324-6. PMID 29187230